CLINICAL TRIAL: NCT05021185
Title: Interactive Mobile Doctor (iMD) to Promote Tobacco Cessation Among Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21727; NCI-2021-09058 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Dependence; Tobacco Use Cessation; Cancer
Keywords: Interactive Mobile Application; Radiation Therapy; Radiation Oncology; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation; Neoplasms; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Mobile Doctor (iMD) Intervention (Experimental): Participants will receive up to a total of 3 iMD sessions prior to their completion of radiation therapy; each session will take about 10-15 minutes and includes: 1) computerized assessments that will be delivered on the screen via text with accompanying audio and participants will respond directly on the tablet 2) tailored videos that deliver messages specific to patient's responses to selected assessment questions and 3) a summary printout
  Interventions: Other: Interactive Mobile Doctor (iMD)
- Control Group (No Intervention): Participants will complete questionnaires and receive a handout containing tobacco cessation resources.

INTERVENTIONS:
Other: Interactive Mobile Doctor (iMD) — Video educational tool
  Arms: Interactive Mobile Doctor (iMD) Intervention

SUMMARY:
The proposed pilot study aims to develop and test a patient video educational tool, an interactive Mobile Doctor (iMD), that can be integrated in radiation oncology setting to effectively engage cancer patients receiving treatment at University of California, San Francisco (UCSF) to facilitate smoking cessation and maintaining smoking abstinence in the context of their radiation treatment.

This study is the first to address tobacco use among can patients receiving radiation therapy that targets both tobacco cessation (current users) and maintaining abstinence (former users who have recently quit).

DETAILED DESCRIPTION:
The interactive Mobile Doctor (iMD) is an interactive video educational program that delivers tailored messages in response to participants' input, generates a summary report providing tobacco use status and cessation resources and solicits participants' interest in receiving referral or information to tobacco cessation resources.

PRIMARY OBJECTIVE:

I. To assess the feasibility and acceptability of the interactive Mobile Doctor (iMD), an interactive patient education tool, utilizing patient-centered and interactive technology approaches to target cancer patients who report using tobacco within the past 12 months and who are receiving or planning to receive radiation therapy for cancer.

SECONDARY OBJECTIVES:

I. To assess preliminary efficacy of iMD on tobacco abstinence when compared to the control (assessment + resource information only).

II. To estimate impacts of iMD on referral requests.

Participants will be randomized to either the iMD or Control Group in a 1:1 ratio, stratified by tobacco use status within past 30 days (current vs former tobacco users), to the iMD intervention or the control group

iMD Intervention Participants: Participants receive up to a total of 3 iMD sessions prior to their completion of radiation therapy (RT). The iMD session will take about 10-15 minutes and will include: 1) computerized assessments(tobacco use in past 12 months and in past 30 days; types of tobacco used, time to first cigarette or tobacco use, cigarettes used per day on a typical day of use, readiness for quitting, and concerns about quitting smoking) that will be delivered on the screen via text with accompanying audio and participants will respond directly on the tablet 2) tailored videos that deliver messages specific to patient's responses to selected assessment questions, including addressing misconceptions of being too late to quit smoking after cancer diagnosis, which could be a barrier for quitting smoking, or tobacco-free is not necessary after completion of RT; and 3) a summary printout, the iMD Summary Reported generated at the end of each iMD session will provide a summary of a participant's RT completion status or anticipated completion date, tobacco use status, plans for quitting or commitment to abstinence, key messages addressing participants' concerns and uniform resource locator (URL)s of the videos watched, California Smokers' Helpline website and telephone numbers, and interest to be contacted by a tobacco treatment specialist or in receiving for tobacco use, referred to tobacco treatment resources.

Control Group Participants: Participants will undergo the assessment questions. Instead of viewing and participating in the interactive video education about tobacco cessation or tobacco-free living, will participants receive a handout containing tobacco cessation resources.

Participants will be followed up for 3 month after their first visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or order
2. Ability to understand study procedures and to comply with them for the entire length of the study.
3. Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
4. Scheduled for a consultation visit with an oncologist to prepare for a radiation therapy for cancer treatment or currently receiving radiation treatment for cancer at a University of California, San Francisco (UCSF) location (Mission Bay, Mount Zion, Parnassus, etc.).
5. Reported using cigarettes, e-cigarette or any tobacco product(s) in the past 12 months

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. Participated in Patient/Care Team Advisory Board Activities for the project
3. Hearing and/or vision disabilities in receiving the iMD intervention or follow-up assessment such as videos or telephone interviews at follow-up
4. Cancer care team's judgement of inappropriateness due to cognitive or medical reasons
5. Inability to understand spoken and written English
6. Completion of radiation therapy for cancer at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible individuals who consent to enroll in the study | Up to 6 months
  The proportion of participants who consent to enroll from the total number who are approached for eligibility will be reported.
Proportion of participants assigned to iMD intervention with a response to referral question | Up to 3 months
  The proportion of participants assigned to iMD intervention who have a recorded response to the question on referral to a smoking cessation treatment service/ resource will be reported.
Proportion of iMD participants who complete 2 or more sessions | Up to 3 months
  The proportion of participants enrolled in the iMD arm who complete at least 2 or more of the iMD sessions will be reported.
Median scores on the perceived helpfulness of the iMD program | Up to 3 months
  The perceived helpfulness of the iMD program will be measured using a 5-point likert scale a a response to the question provided to the participants who are assigned to the iMD arm which rates the helpfulness of the intervention as 1='Somewhat helpful" to 5="Very helpful

SECONDARY OUTCOMES:
Proportions of participants with reported abstinence | Up to 3 months
  Proportions of participants with self-report + biochemically verified tobacco abstinence (salivary cotinine or exhaled CO)
Proportion of iMD participants who indicate requests of referral for smoking cessation | Up to 9 months
  The investigators will estimate impacts of iMD on yield referral requests (when participants respond "Yes" to be referred for smoking cessation related services) for participants assigned to the iMD program

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No